CLINICAL TRIAL: NCT02137174
Title: The Efficacy of Constructed Intervention by Home and School Visits on Glycemic Control in Children With Type I Diabetes
Brief Title: Home and School Visits Intervention for Children With DM TYPE 1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Eli Hershkovitz, Head of Pediatric Endocrinology Unit, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EH-diab013
Record Dates: First submitted 2014-05-10; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home and school visits (Active Comparator)
  Interventions: Other: Home and school visits
- Control (No Intervention)

INTERVENTIONS:
Other: Home and school visits — Each child in the intervention group received, in addition to the standard care at the diabetic clinic, home and school visits by a multidisciplinary team during one year.
  Arms: Home and school visits

SUMMARY:
Home and school visits by multidisciplinary team will improve metabolic control in kids having insulin dependent diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* HbA1c ≥ 8% at baseline, and diabetes duration of at least 7 months.

Exclusion Criteria:

* Patients during honeymoon period
* Patients and their parents who do not speak Hebrew or Arabic
* Patients who were not under any educational system
* Patients who had other severe chronic disorders

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
HBA1C | 2 YEARS

SECONDARY OUTCOMES:
Number of DKA episodes | 2 YEARS
Number of Hospitalizations | 2 years
Hypoglycemia rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Endocrinology Unit, Soroka Medical Center, Beersheba, Israel